CLINICAL TRIAL: NCT04867109
Title: Multicenter Prospective Study Evaluating the Interest of HE4 in the Diagnostic Approach of Endometrial Cancer in Patients With Postmenopausal Bleeding
Brief Title: HE4 in the Diagnostic Approach of Endometrial Cancer in Patients With Postmenopausal Bleeding
Acronym: METRODEC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nantes University Hospital (Other)
Collaborators: Roche Diagnostics GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: RC21_0166
Record Dates: First submitted 2021-04-13; First posted 2021-04-30 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Endometrial Neoplasms; Postmenopause; Uterine Hemorrhage; Cancer Biomarker; CA 125 Antigen
Keywords: Endometrial cancer; Human epididymis protein 4; HE4; CA125; Post-menopausal bleeding
MeSH Terms: conditions — Endometrial Neoplasms; Uterine Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Patients with Post menopausal bleeding — Any patient presenting post-menopausal bleeding who is to undergo hysteroscopy or hysterectomy will have an additional blood tube taken during her pre-operative blood work-up for the determination of the serum markers HE4 and CA125, after having obtained her non-opposition to participate in the study.
  The blood tube collected for the research will be sent to the biochemistry laboratory of the Nantes University Hospital for a centralized analysis.
  This analysis will be done sequentially and the results will not be transmitted to the investigator.
  At D0, the day of surgery, the operative report will be retrieved as well as the quality of life questionnaires SF12 and PGI-I and the acceptability questionnaire completed before surgery.
  At 1 month after surgery, the anatomopathological results will be retrieved as well as the value of the tumour markers CA125 and HE4.
Diagnostic Test: CA125 and HE4 assays — Blood was collected in a standard heparinized vial. Samples were sent to a central laboratory unit (biochemistry laboratory at the Nantes university hospital), centrifuged and plasmas were stored at -20°C until analysis. Plasma CA125 and HE4 concentrations were determined by run in single measurements using an electrochemiluminescence Elecsys immunoassay (ECLIA) on a Roche Diagnostics Cobas 8000® e602 analyser (Roche Diagnostics, Mannheim, Germany).

SUMMARY:
This study aims to explore the sensitivity of an innovative marker, HE4, in the diagnosis approach of endometrial cancer in case of postmenopausal bleedings.

DETAILED DESCRIPTION:
Endometrial cancer is the most common pelvic gynecological cancer in France, ranking 5th among cancers in women in terms of incidence.

The most frequent symptom is post-menopausal bleeding and is one of the primary reasons for consultation in gynecological emergencies.

The diagnosis of endometrial cancer is made by histological analysis of endometrial tissue taken during a surgical intervention. The latter is mostly reassuring.

These interventions are often performed in mild situations and there is currently no element to be sufficiently reassuring to avoid surgery.

At present, there is no biological marker used in current practice. In the population of patients with post-menopausal bleeding requiring surgical exploration for diagnosis, the pathology results are often reassuring. These procedures could have been avoided, especially as these patients often have numerous co-morbidities and these surgeries are therefore more risky. The appearance of a new tumour marker could be useful in the management of these patients and avoid many unnecessary and risky surgeries

This study aims to explore the sensitivity of an innovative marker, HE4, in the diagnosis approach of endometrial cancer in case of postmenopausal bleedings.

ELIGIBILITY:
Inclusion Criteria:

* Patient with postmenopausal bleeding
* Patient requiring hysteroscopy or hysterectomy
* No objection from the patient to participate in the study

Exclusion Criteria:

* Non-menopausal patient
* Patient under guardianship, curatorship or deprived of her freedom
* Patient with proven metastases on imaging
* Patient with a macroscopically suspicious cervix
* Patient presenting an ovarian cyst or an associated adnexal pathology
* Patient contraindicated for surgical treatment (therefore not eligible for pathological analysis)
* Patient who has already been treated with hormone therapy for breast cancer
* Patient who has already had surgery for this pathology, with a contributing anatomopathological result (we will therefore include patients who would not benefit from an operative hysteroscopy after performing a cornier® pipelle that does not allow a positive result)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Adults women
Study Population: Any patient with postmenopausal bleeding who is to undergo hysteroscopy or hysterectomy will have an additional blood tube taken during her pre-operative blood work-up for the measurement of the serum markers HE4 and CA125 after she has indicated that she does not wish to participate in the study
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-06-25 (Actual); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate the sensitivity of the HE4 marker in patients with postmenopausal bleeding in the diagnosis of endometrial cancer | Until the pathological results (About 10-15 days)
  The HE4 assays will be performed using the electrochemiluminescence (ECL) technique on Cobas Pro module E801, Roche Diagnostics. The HE4 assay is based on a sandwich-type electrochemiluminescence method. The HE4 assay with the Roche Diagnostics Elecsys reagent has been standardized against the Fujirebo Diagnostics HE4 EIA method.
  Positive/negative HE4 result for the estimation of the sensitivity of HE4 in the diagnosis of endometrial cancer.
  The commonly accepted threshold for ovarian cancer management of 140pmol/l in postmenopausal patients should be used.
  The gold standard for endometrial cancer is the pathological result (absence/presence of cancer) of the sample taken.

SECONDARY OUTCOMES:
Assess other diagnostic parameters (specificity, PPV, NPV) of HE4 | Until the pathological results (About 10-15 days)
  ROC curve for the HE4 marker in the diagnosis of endometrial cancer.
Establish the optimal threshold of HE4 for the diagnosis of endometrial cancer (use of an ROC curve) | Until the pathological results (About 10-15 days)
  Search for the threshold with the best specificity of HE4 in the diagnosis of endometrial cancer
Evaluate the diagnostic capabilities of CA125 alone and in combination with HE4, as well as the REM and REM-B algorithms for the diagnosis of endometrial cancer | Until the pathological results (About 10-15 days)
  Estimation of sensitivity, specificity, PPV and NPV in the diagnosis of endometrial cancer for the CA125 biomarker and the REM and REM B algorithms
Establish the existence of thresholds for HE4 and/or CA125 markers predictive of disease severity (FIGO stage) | Until the results of the extension assessment in the event of proven endometrial cancer (1 month)
  Search for HE4 and CA125 marker thresholds to assess disease severity by FIGO stage
Reassess the pathological threshold value of endometrial thickness on ultrasound | Until the pathological results (About 10-15 days)
  Search for the pathological threshold of endometrial thickness in the diagnosis of endometrial cancer
Assess the relationship between endometrial thickness on ultrasound and HE4 and CA125 marker values | Until the pathological results (About 10-15 days)
  Estimation of the relationship between CA125 and HE4 markers and endometrial thickness on ultrasound
To evaluate the diagnostic capabilities of HE4 and CA125 in subgroups of smoking patients and patients with renal failure | Until the pathological results (About 10-15 days)
  Estimation of sensitivity, specificity, PPV and NPV in the diagnosis of endometrial cancer for HE4 and CA125 in patients with active smoking and/or renal failure
Identify potential confounding factors associated with the value of the HE4 marker like treatments, comorbidities (renal insufficiency, high BMI) and others criteria that are collected in the medical files | Until the pathological results (About 10-15 days)
  Analyses of variables measured at inclusion that may influence the value of the HE4 marker.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Saint-Nazaire Hospital, Saint-Nazaire, Loire-Atlantique
  - Vendee Hospital Center, La Roche-sur-Yon, Vendee

IPD SHARING:
Plan to Share IPD: No